CLINICAL TRIAL: NCT00151645
Title: Renal Cell Carcinoma Treatment With Activated Tumor- Infiltrated Lymphocytes. A Non-Randomized Phase II Trial.
Brief Title: Efficacy of Activated Lymphocytes in Renal Cell Carcinoma.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFSSAPS 990434; PHRC/02-06; CIC0203/013
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2006-01-02 (Estimated); Status verified 2005-12

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Immunotherapy; Renal cell carcinoma; Metastasis; Lymphokine activated killers; Cell therapy
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — CD83 protein, human

INTERVENTIONS:
Drug: activated lymphocytes

SUMMARY:
Renal cell carcinoma represents today 3% of the solid tumors of the adult. Their bad prognosis is due to the frequency of metastasis and the resistance to chemotherapy. Immunotherapy (interferon-α, interleukin-2) has shown some good results but an important toxicity. In our study, we evaluate the response to a new therapeutic strategy which combines an injection of patient's own activated lymphocytes to a classic immunotherapy with interferon-α and interleukin-2.

DETAILED DESCRIPTION:
Phase I and II trials for the treatment of melanoma or renal cell carcinoma have already evaluated lymphokine-activated killer cells and tumor-infiltrating cells. In metastatic renal cell carcinoma, these therapies have shown some complete responses and a low toxicity. In our study, we evaluate the response to a new therapeutic strategy which combines an injection of patient's own activated lymphocytes to a classic immunotherapy with interferon-α and interleukin-2. A secondary objective is to improve cell preparation methods and to characterize functionally and phenotypically injected cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years
* Metastatic renal adenocarcinoma histologically proven
* Karnofsky performance status ≥ 70%
* Life expectation > 3 months
* At least one target, in a non-irradiated area
* Objective response or steady-state after a treatment with cytokines
* Informed written consent

Exclusion Criteria:

* Patients presenting more than one metastatic site with one hepatic metastasis diagnosed within the last 12 months
* White blood cells count < 2.5 G/L, Platelet count < 100 G/L
* Serum creatinine rate > 150 µmol/L
* Positive serology for : hepatitis B, hepatitis C, retrovirus
* Patient not available for a long-term follow-up
* Bellini duct tumor
* History of allograft or tumor within the five past years
* Severe cardiovascular, hepatic, renal or pulmonary troubles
* Auto-immune disease
* Severe infection
* Pregnancy or breast-feeding
* Corticotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2003-12; Study Completion 2005-07

PRIMARY OUTCOMES:
Objective response rate: partial or complete response during at least 4 weeks from week 22 after the beginning of the first cycle of cytokines.

SECONDARY OUTCOMES:
- Disease free survival
- Overall survival
- Functional and phenotypic characteristics of injected cells
- Biological response

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Catros-Quemener, PharmD, PhD, Study Director — CHU Rennes; Eric Bellissant, MD, PhD, Study Chair — CHU Rennes; François Guillé, MD, Principal Investigator — CHU Rennes
Locations (1):
- Service d'Urologie - Hôpital Pontchaillou, Rennes, France

REFERENCES:
- [Background] Belldegrun A, Pierce W, Kaboo R, Tso CL, Shau H, Turcillo P, Moldawer N, Golub S, deKernion J, Figlin R. Interferon-alpha primed tumor-infiltrating lymphocytes combined with interleukin-2 and interferon-alpha as therapy for metastatic renal cell carcinoma. J Urol. 1993 Nov;150(5 Pt 1):1384-90. doi: 10.1016/s0022-5347(17)35785-3. PMID 8411405
- [Background] Figlin RA, Pierce WC, Kaboo R, Tso CL, Moldawer N, Gitlitz B, deKernion J, Belldegrun A. Treatment of metastatic renal cell carcinoma with nephrectomy, interleukin-2 and cytokine-primed or CD8(+) selected tumor infiltrating lymphocytes from primary tumor. J Urol. 1997 Sep;158(3 Pt 1):740-5. doi: 10.1097/00005392-199709000-00012. PMID 9258071
- [Background] Hayakawa M, Hatano T, Ogawa Y, Gakiya M, Ogura H, Osawa A. Treatment of advanced renal cell carcinoma using regional arterial administration of lymphokine-activated killer cells in combination with low doses of rIL-2. Urol Int. 1994;53(3):117-24. doi: 10.1159/000282651. PMID 7645136
- [Background] Mathiot C, Thiounn N, Tartour E, Flam T, Peyret C, Joyeux I, Zerbib M, Brandely M, Debre B, Fridman WH. Non-cytotoxic CD4 tumour-infiltrating lymphocytes induce responses in patients with metastatic renal cell carcinoma previously treated with interleukin-2. Eur J Cancer. 1995;31A(9):1551-2. doi: 10.1016/0959-8049(95)00235-b. No abstract available. PMID 7577091